CLINICAL TRIAL: NCT07019246
Title: Safety of Etomidate-propofol Mixture vs. Propofol for Total Intravenous Anesthesia in Elderly Patients Undergoing Abdominal Surgery - A Randomized, Double-blind, Controlled Study
Brief Title: Safety of Etomidate-propofol Mixture vs. Propofol for Total Intravenous Anesthesia in Elderly Patients Undergoing Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shiyong Li, Associate Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEPTE
Record Dates: First submitted 2025-05-16; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Etomidate Combined With Propofol; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP group (Experimental): Patients in this group will receive etomidate- propofol mixture during induction and maintenance.
  Interventions: Drug: EP mixture
- P group (Active Comparator): Patients in this group will receive propofol during induction and maintenance.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: EP mixture — Patients will receive etomidate - propofol mixture during induction and maintenance. Sufentanil 0.2-0.7 μg/kg，Cisatracurium 0.15 mg/kg，EP mixture（E：P=1:2） 0.1-0.25 ml/kg for induction, EP mixture 0.4~ 1.2 ml/kg/h and remifentanil 0.05μg/kg/min ~0.3 μg/kg/min for maintenance.
  Arms: EP group
Drug: Propofol — Patients will receive propofol during induction and maintenance.Sufentanil 0.2-0.7 μg/kg，Cisatracurium 0.15 mg/kg，propofol 0.1-0.25 ml/kg for induction, propofol 0.4~ 1.2 ml/kg/h and remifentanil 0.05μg/kg/min ~0.3 μg/kg/min for maintenance.
  Arms: P group

SUMMARY:
The purpose of this study is to access the safety of etomidate - propofol mixture vs propofol for total intravenous anesthesia in elderly patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is one of the commonly used methods for maintaining anesthesia in clinical practice. The commonly used intravenous anesthetic drugs in clinical settings include propofol and etomidate. Both have their own advantages and disadvantages in clinical application. Among them, propofol has the advantages of rapid onset, complete sedation, and quick awakening, but it is prone to injection pain, and its inhibitory effect on the circulatory system is relatively significant. The incidence of hypotension during TIVA surgery with propofol is relatively high; while hypotension during surgery significantly increases the risk of adverse cardiovascular events during the perioperative period. Etomidate is a derivative of imidazole, and it can increase the reversibility of GABAA receptor activity, inhibit synaptic transmission and impulse conduction, and exert a sedative effect. Etomidate has a rapid onset, has a minor impact on hemodynamics, and has a shorter time-quantity-related half-life compared to propofol. However, etomidate has an inhibitory effect on the adrenal cortex. Numerous studies have confirmed that etomidate, when administered as a single injection or continuous infusion, can temporarily inhibit the function of the adrenal cortex, and the adrenal cortex function of patients can recover to the preoperative baseline level within 48 hours after surgery .

Comprehensive drug administration can reduce adverse reactions caused by a single drug. Considering the complementary pharmacodynamic effects of propofol and etomidate, the combination of the two drugs is beneficial for maximizing their respective advantages and reducing adverse reactions. In vitro drug tests have confirmed that the mixture of etomidate and propofol has physical and chemical compatibility for up to 24 hours at refrigerated temperature (4℃), room temperature (25℃), and body temperature (37℃), which creates the prerequisite conditions for the mixed use of propofol and etomidate.

The etomidate-propofol mixture is currently widely used for sedation during colonoscopy, gastroscopy, and bronchoscopy, providing a complete sedative effect, and the advantages of the mixed use have been observed, such as a low incidence of hypotension after administration, low incidence of injection pain and muscle tremors, and a low incidence of nausea and vomiting after awakening . The etomidate-propofol mixture is used for TIVA in most small-sample observational studies. A prospective observational study found that the etomidate-propofol mixture has a definite clinical efficacy for elderly patients undergoing spinal surgery, with a lower incidence of hypotension, reduced cerebral oxygen metabolism, reduced postoperative neurological complications, and no increase in the incidence of drug adverse reactions . However, there is a lack of research on the safety of the etomidate-propofol mixture for other elderly surgeries during general anesthesia maintenance.

Hypotension during surgery is a common complication during general anesthesia. Severe hypotension is closely related to perioperative cardiovascular complications and stroke . Elderly patients have a higher risk during the perioperative period. Therefore, avoiding perioperative hypotension is a basic prerequisite for ensuring patient safety. Abdominal surgery is a common type of general surgery, with a large number of surgeries and relatively consistent operation times, making it convenient for case collection. Therefore, in elderly patients scheduled for elective abdominal surgery, this study explores the impact of the propofol-etomidate mixture on the incidence of hypotension during anesthesia induction and maintenance, with the aim of providing a selectable, safe, reasonable, and easily scalable medication regimen for elderly patients undergoing total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ~Ⅲ;
* BMI was 18-28 kg/m2;
* For elective abdominal surgery under intravenous general anesthesia;
* The expected duration of anesthesia was 1 to 4 hours.

Exclusion Criteria:

* Septic shock and multiple organ failure diagnosed within 14 days;
* Hyperkalemia (serum potassium >5.5mmol/L) within 48 hours;
* Stroke or transient ischemic attack within 3 months;
* Patients with unstable angina pectoris or myocardial infarction within 3 months; Arrhythmia requiring treatment was not treated or treatment did not meet expectations;
* Patients with preoperative diagnosed diabetes mellitus and uncontrolled blood glucose; Diabetic complications were diagnosed before surgery, including diabetic ketoacidosis, hyperosmolar coma, diabetes-related infection, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot, etc.
* Severe liver and renal dysfunction;
* Liver surgery, renal surgery, adrenal surgery, day surgery;
* Resting blood pressure ≥180/110 mmHg (2020 ISH hypertension guideline ≥ grade 3 hypertension); Or systolic blood pressure <90mmHg or mean blood pressure <65mmHg.
* Taking corticosteroids or other immunosuppressants for more than 10 days within 6 months or having a history of adrenal cortex suppression or immune system diseases;

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and duration of hypotension during anesthesia | day 1 (The time from the start of anesthesia induction to extubation)
  Blood pressure fluctuations greater than 10% relative to baseline values

SECONDARY OUTCOMES:
Success rate of sedation | day 1 (The time from the start of anesthesia induction to extubation)
  ① Successful induction of anesthesia, MOAA/S score to 0 or BIS<60 within 3 minutes after the end of administration; ② During the maintenance of anesthesia, there was no single BIS>60 for more than 5 minutes or the cumulative BIS>60 for more than 20% of the anesthesia time, no anticipated limb movement, and no anesthesia rescue measures during the maintenance period
Recovery time | Day 1 (Time from drug withdrawal to extubation)
  Time from drug withdrawal to extubation
The type and dosage of vasoactive drugs used during operation | day 1 (The time from the start of anesthesia induction to extubation)
  The type and dosage of vasoactive drugs used during operation
The incidence of postoperative nausea and vomiting | within 72 hours after surgery
  The severity of postoperative nausea and vomiting is evaluated using a Numerical Rating Scale（NRS）.Patients select a number to indicate nausea/vomiting severity:0 for none,1 -3 for mild,4-6 for moderate, and 7-10 for severe.
The incidence of in-hospital complications after surgery | Perioperative
  Complications in the cardiovascular, respiratory, renal and other systems that occurred in the hospital Complications in the cardiovascular, respiratory, renal and other systems that occurred in the hospital after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shiyong Li, Principal Investigator — Department of Anesthesiology of Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No